CLINICAL TRIAL: NCT01208532
Title: Quality of Life in Patients With Stem Cell Transplant After High Dose Chemotherapy: Validation Study of the Korean Version of the EORTC QLQ-HDC29
Brief Title: Validation Study of the Korean Version of the EORTC QLQ-HDC29
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sung-Soo Yoon, Professor, Seoul National University Hospital
Other Study IDs: HDC29_Kor
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Quality of Life After Stem Cell Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to evaluate the reliability and validity of the Korean version of the European Organization for Research and Treatment of Cancer High-dose Chemotherapy module (EORTC HDC-29).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are aged more than 18 years
* Patients who are diagnosed with hematologic malignancies and who are planned to receive high-dose chemotherapy followed by allogeneic or autologous stem cell transplantation (SCT)
* Patients who agree with the informed consent

Exclusion Criteria:

* Patients who are unable to complete the questionnaire due to the serious physical or psychological morbidity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are diagnosed with hematologic malignancies and who are planned to recieve high-dose chemotherapy followed by allo or auto stem cell transplantation in Seoul National University Hospital, Korea
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2010-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Reliability and validity of the Korean version of the EORTC HDC-29 | at the patient's hospitalization (before the SCT) and the outpatient clinic (three, six, and 12 months after their SCT)
  Relaibility; Cronbach's alpha coefficient is used to evaluate the internal consistency.
  Validity; Persons's correlation coefficient is used to examine the correlation between similar dimensions of the different questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Soo Yoon, MD, PhD, Principal Investigator — Seoul National University Hospital; Jung Mi Oh, Pharm.D., Principal Investigator — College of Pharmacy, Seoul National University
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Velikova G, Weis J, Hjermstad MJ, Kopp M, Morris P, Watson M, Sezer O; EORTC Quality of Life Group. The EORTC QLQ-HDC29: a supplementary module assessing the quality of life during and after high-dose chemotherapy and stem cell transplantation. Eur J Cancer. 2007 Jan;43(1):87-94. doi: 10.1016/j.ejca.2006.09.004. Epub 2006 Nov 1. PMID 17081744
- [Background] Yun YH, Park YS, Lee ES, Bang SM, Heo DS, Park SY, You CH, West K. Validation of the Korean version of the EORTC QLQ-C30. Qual Life Res. 2004 May;13(4):863-8. doi: 10.1023/B:QURE.0000021692.81214.70. PMID 15129896
- [Background] Han CW, Lee EJ, Iwaya T, Kataoka H, Kohzuki M. Development of the Korean version of Short-Form 36-Item Health Survey: health related QOL of healthy elderly people and elderly patients in Korea. Tohoku J Exp Med. 2004 Jul;203(3):189-94. doi: 10.1620/tjem.203.189. PMID 15240928
- [Background] Yoo H, Lee K, Lee J, Eremenco S, Choi S, Kim H, Lee J. Korean translation and validity of FACT-BMT version 4 and the quality of life in allogeneic bone marrow transplantation patients. Qual Life Res. 2006 Apr;15(3):559-64. doi: 10.1007/s11136-005-1769-3. PMID 16547794